CLINICAL TRIAL: NCT04308135
Title: The Clinical and Neuroimaging Differences Between Patients With Vascular Parkinsonism and Idiopathic Parkinson's Disease
Brief Title: Differences Between Patients With Vascular Parkinsonism and Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ali Shalash, professor of Neurology, Ain Shams University
Other Study IDs: MD209/2019
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Vascular Parkinsonism; Parkinson's Disease
Keywords: Parkinson's Disease; vascular parkinsonism; MRI brain; non-motor
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples for biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- vascular parkinsonism: the investigators will recruit 30 patients diagnosed as Vascular Parkisonism ,
  Interventions: Diagnostic Test: Neuro-radiological tools:; Diagnostic Test: cognitive tests; Diagnostic Test: lab investigations; Diagnostic Test: Beck depression inventory (BDI)(Arabic version); Diagnostic Test: Clinical Tools for Urinary symptoms:; Diagnostic Test: Freezing of gait questionnaire; Diagnostic Test: non-motor symptoms scales (NMSS).; Diagnostic Test: Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS):; Diagnostic Test: ELIZA for alpha-synuclein; Other: transcranial color-coded duplex(TCCD); Other: extracranial carotid duplex; Other: The Arabic version of Parkinson's Disease Questionnaire( PDQ-39)
- Parkinson's disease: 50 patients diagnosed as Parkinson Disease
  Interventions: Diagnostic Test: Neuro-radiological tools:; Diagnostic Test: cognitive tests; Diagnostic Test: lab investigations; Diagnostic Test: Beck depression inventory (BDI)(Arabic version); Diagnostic Test: Clinical Tools for Urinary symptoms:; Diagnostic Test: Freezing of gait questionnaire; Diagnostic Test: non-motor symptoms scales (NMSS).; Diagnostic Test: Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS):; Diagnostic Test: ELIZA for alpha-synuclein; Other: transcranial color-coded duplex(TCCD); Other: extracranial carotid duplex; Other: The Arabic version of Parkinson's Disease Questionnaire( PDQ-39)
- Controls: 30 healthy controls.
  Interventions: Diagnostic Test: cognitive tests; Diagnostic Test: Beck depression inventory (BDI)(Arabic version); Diagnostic Test: Clinical Tools for Urinary symptoms:; Diagnostic Test: Freezing of gait questionnaire; Diagnostic Test: non-motor symptoms scales (NMSS).; Diagnostic Test: Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS):; Other: transcranial color-coded duplex(TCCD); Other: extracranial carotid duplex; Other: The Arabic version of Parkinson's Disease Questionnaire( PDQ-39)

INTERVENTIONS:
Diagnostic Test: Neuro-radiological tools: — MRI brain: to measure white matter
  c) Ultrasonographic examination of extracranial vessels: The intimal medial thickness of the common carotid artery (CCA-IMT) will be measured in B-mode. The carotid arteries will be evaluated for the presence of atherosclerotic lesions (plaques) either soft or hard .The residual lumen and degree of stenosis will be measured. The peak systolic velocity will be detected.
  Other Names: magnetic resonance imaging (MRI)
  Groups: Parkinson's disease; vascular parkinsonism
Diagnostic Test: cognitive tests — All patients will be evaluated for global cognitive assessment by: Montreal Cognitive Assessment (MoCA) (Arabic version) Visuospatial skills will be assessed by Clock Drawing Tests from MoCA test and copy the intersecting pentagons from Addenbrooke's test (Arabic version) Language will be examined by semantic fluency from Addenbrooke's test (Arabic version) and similarities from Wechsler Adult Intelligence Scale (WAIS) Attention will be evaluated by digit span from Wechsler test),and by the number of seconds needed to sequence numbers using a pencil (Trail making test A) from MoCA test . For the evaluation of memory, participants will complete Wechsler memory subset
  , and the investigators also will use their three-item recall from the Mini-Mental State Examination( MMSE). Executive functions will be measured by Wisconsin card sorting test and also verbal fluency test from Addenbrooke's test. Frontal Assessment Battery (FAB) scale
Diagnostic Test: lab investigations — Each patient will undergo full lab investigations:[lipid profile ,complete blood count, uric acid ,Hemoglobin A1c (HbA1c), liver functions, renal functions, and electrolytes]
  Groups: Parkinson's disease; vascular parkinsonism
Diagnostic Test: Beck depression inventory (BDI)(Arabic version) — Clinical Tool for depression
Diagnostic Test: Clinical Tools for Urinary symptoms: — the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) Scale (Arabic version)
Diagnostic Test: Freezing of gait questionnaire — Clinical Tools for Gait (in on and off state ), Gait will be assessed by:
  * .Freezing of gait questionnaire
  * Berg balance scale.
  * 10 meter walk test .
  * Timed up and go test.
Diagnostic Test: non-motor symptoms scales (NMSS). — Clinical Tool for assessment of non-motor symptoms of PD
Diagnostic Test: Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS): — Clinical Tools for assessment of the neurological severity and stage of disease Clinical Tool for assessment of the neurological severity and stage of disease during "OFF" and "ON" states, Hoehn and Yahr scale. The presence of lower limb parkinsonism will be determined by a two-point difference between upper limb and lower limb scores of bradykinesia, rigidity or postural instability from part III of the MDS-UPDRS. Patients will be examined in the early morning, in 'OFF' state, with MDS-UPDRS, Hoehn and Yahr and freezing of gait questionnaire(FOG-Q) scales. Immediately afterwards, they will take their regular first dose of levodopa. After 1 hour, patients will be examined again with the same tests and scales.
  Response to levodopa will be determined as patients who reached a percentage reduction exceeding 25% in part III of the MDS-UPDRS
Diagnostic Test: ELIZA for alpha-synuclein — measuring serum of alpha-synuclein, tau and their autoantibodoies
  Groups: Parkinson's disease; vascular parkinsonism
Other: transcranial color-coded duplex(TCCD) — TCCD using phase array 2.4 Hz probe for evaluation of cerebral vasomotor reactivity (CVR) by measuring the Breath holding index(BHI),flow velocities and pulsatility index of middle cerebral artery and posterior cerebral artery on both sides.
Other: extracranial carotid duplex — to assess atherosclerosis, stenosis of carotids
Other: The Arabic version of Parkinson's Disease Questionnaire( PDQ-39) — Clinical tool for quality of life of PD patients

SUMMARY:
Vascular parkinsonism (VP) is defined as the presence of parkinsonian syndrome, evidence of cerebrovascular disease by brain imaging and an established relationship between the two disorders.

However, the diagnosis of VP is problematic. This study aims to distinguish VP from Parkinson's disease (PD) in multiple aspects including clinical features as motor ,non motor symptoms

,response to treatment ,cognitive assessments by using multiple scales, neuro-radiological features of magnetic resonance imaging (MRI) and transcranial color-coded duplex (TCCD) findings. This differentiation will have therapeutic and prognostic implications .

DETAILED DESCRIPTION:
Type of Study : case -control comparative study.

• Study Setting: Patients with VP and patients with PD from movement disorders and stroke outpatient clinics in Ain shams University Hospitals.

Sampling Method study of consecutive patients in Ain Shams University clinic, who had been regularly followed up in the clinic and already had a diagnosis either VP or PD at the time of data collection.

Sample Size: 30 patients diagnosed as VP, 50 patients diagnosed as PD, and 30 healthy age and sex matched controls. The difference in selected quantitative variables used to evaluate the participants is used to estimate the sample size.

This study aims to distinguish VP from Parkinson's disease(PD) in multiple aspects including clinical features as motor ,non-motor symptoms, response to treatment ,cognitive assessments by using multiple scales, neuro-radiological features of magnetic resonance imaging (MRI) and transcranial color-coded duplex(TCCD)findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD or VP, and healthy controls will be included in the study.
* PD diagnosis will be based on the Queen Square Brain Bank for Neurological Disorders clinical criteria and MDS criteria.
* The VP patients will be included if they fulfill the following criteria (Zijlman's diagnostic criteria)Parkinsonism presentation (at least two of the cardinal features: tremors, bradykinesia, rigidity and postural instability).

Cerebrovascular disease, defined as evidence of relevant cerebrovascular disease by brain imaging or the presence of focal signs or symptoms consistent with stroke.

A relationship between (1) and (2): acute or delayed progressive onset of parkinsonism.

Based on the above criteria, two forms of VP are suggested: one with acute onset, and another one with insidious progression. The diagnosis will be confirmed by assigning a vascular score. Two points or more are essential to diagnose VP. The points will be assigned as follows:

* Two points: Pathologically or angiographically proven diffuse vascular disease.
* One point: Onset of parkinsonism within 1 month of clinical stroke.
* One point: History of two or more strokes.
* One point: Neuroimaging evidence of vascular disease in two or more vascular territories.
* One point: History of two or more risk factors for stroke (hypertension, smoking, diabetes mellitus, hyperlipidaemia, presence of heart disease associated with stroke [coronary artery disease, atrial fibrillation, congestive heart failure, valvular heart disease, mitral valve prolapse, and other arrhythmias], family history of stroke, history of gout, and peripheral vascular disease)

Exclusion Criteria:

* PD patients with age at onset less than 40 years.
* Any alternative cause that significantly impair gait.
* Inability of the patient to undergo neuroimaging.
* Patients couldn't perform the test or severely demented.
* Atypical and other secondary parkinsonism as patients who had a history of toxin exposure.or antipsychotic drugs treatment by history ,neurological examination and brain MRI .
* Family or patient's refusal to give written consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 30 patients diagnosed as VP, 50 patients diagnosed as PD
  , and 30 healthy age and sex matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
MDS-UPDRS scale on on and off state | 2 year... will be at single point
  It detects the motor differences between Vascular Parkinsonism and Parkinson's Disease by scores on the scale ...the maxium score is 199 represents the worst (total disability) with a score of zero representing (no disability)
Montreal Cognitive Assessment (MoCA) (Arabic version) | 2 years....will be at single point
  MoCA scores range between 0 and 30. .high score more than or equal 26 is normal
White matter severity by MRI brain | 2 years....will be at single point
  White matter differences by fazekas scale 0,1,2 or 3 scores
Non motor symptoms scale | 2 years.....will be at single point
  It detects the non motor symptoms differences between Vascular Parkinsonism and Parkinson's Disease byUsing a distribution of NMSS scores by quartiles, a classification based on levels from 0 (no NMS at all) to 4 (very severe NMS) for 30 itemes ...high score is worst
Addenbrooke's test (Arabic version) | 2 year ....will be at single point
  for aassement of Visuospatial skills, Language and verbal fluency result score 16 for visuospatial processing ,26 for language 14 for fluency high score is best
Wechsler Adult Intelligence Scale (WAIS) | 2 year....will be at single point
  The average score for the test is 100, and any score from 90 to 109 is considered to be in the average intelligence range. Score from 110 to 119 are considered to be High Average. Superior scores range from 120 to 129 and anything over 130 is considered Very Superior.
Frontal Assessment Battery scale. | 2 year ....will be at single point
  Frontal Assessment Battery scale..total score is from a maximum of 18, higher scores indicating better performance.

SECONDARY OUTCOMES:
Substantia nigra Echogenicity by transcranial doppler | 2 years
  to detect differences of substantia nigra Echogenicity by millimeter and differences of mean flow velocities by centimeter per second
Carotid arties wall thickness by Extra cranial duplex | 2 year
  to detect differences of Intima-media thickness values by millimeter and flow velocities by centimeter per second

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] George P, Roushdy T, Fathy M, Hamid E, Ibrahim YA, El-Belkimy M, Abdulghani MO, Shalash A. The clinical and neuroimaging differences between vascular parkinsonism and Parkinson's disease: a case-control study. BMC Neurol. 2024 Feb 6;24(1):56. doi: 10.1186/s12883-024-03556-9. PMID 38321372